CLINICAL TRIAL: NCT07313475
Title: Evaluation of the Cryocheck HexLA Integrated TCA for the Detection of Lupus Anticoagulant
Acronym: HEXLA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9486
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lupus Anticoagulant
Keywords: Lupus Anticoagulant; Coagulation; Phospholipid; Time activated partial thromboplastin (TCA); Cryocheck HexLA; Cephen LS
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lupus anticoagulant (LA) testing is performed using two screening tests: activated partial thromboplastin time (APTT) and diluted Russell's viper venom time. If one of the screening tests is positive, a confirmation test based on the same principle is performed.

The HUS Hematology Laboratory uses an integrated APTT for LA testing, consisting of a screening reagent: Cephen LS, and a confirmation reagent: Cephen (Hyphen Biomed).

The aim of this study is to determine whether another integrated activated partial thromboplastin time (APTT) test, Cryocheck HexLA, offers better performance than Cephen LS/Cephen, both in terms of sensitivity to lupus anticoagulant (LA) and susceptibility to interference from anticoagulant treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (≥ 18 years)
* Sample sent to the HUS Hematology Laboratory and analyzed for LA detection as part of routine care.

Exclusion Criteria:

- Insufficient sample volume

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject blood sample already analyzed in the laboratory as part of the treatment by the reference method
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Cryocheck HexLA compared to Cephen LS/Cephen reagents with regard to lupus anticoagulant (LA) | Up to 9 months
  A Fisher or McNemar statistical test on paired samples will be performed by comparing the results (positive or negative) of the integrated Cephen LS/Cephen and Cryocheck HexLA TCA tests, performed on the same sample, in patients not receiving anticoagulant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - CHU de Strasbourg - France, Strasbourg, France